CLINICAL TRIAL: NCT01887197
Title: Repeatability and Response Study of Absorptive Clearance Scans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tim Corcoran (Other)
Responsible Party: Sponsor-Investigator, Tim Corcoran, PhD, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1RO1 HL108929-01 (B); 1R01HL108929-01 (NIH)
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-06

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; mucociliary clearance; airway surface liquid; nuclear medicine; mannitol
MeSH Terms: conditions — Cystic Fibrosis | interventions — Mannitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Repeatability (Experimental): Subjects perform two sequential absorptive clearance scans (within 30 days) to determine the repeatability of the technique. Subjects also perform a third scan two years later so that longitudinal change can be measured.
  Interventions: Other: Absorptive clearance scan
- Response (Experimental): Subjects perform three different absorptive clearance scans. One is a baseline measurement while the other two measure absorptive clearance after an intervention (inhaled hypertonic saline, mannitol inhalation powder).
  Interventions: Other: Absorptive clearance scan; Drug: inhaled hypertonic saline (7%); Drug: mannitol inhalation powder

INTERVENTIONS:
Other: Absorptive clearance scan — Subjects inhale a nebulized mixture of the radiopharmaceuticals Indium 111-DTPA and Technetium 99m sulfur colloid.
Drug: inhaled hypertonic saline (7%) — nebulized hypertonic saline (7%)
  Other Names: Hypersal
  Arms: Response
Drug: mannitol inhalation powder — mannitol inhalation powder
  Other Names: Bronchitol
  Arms: Response

SUMMARY:
The investigators are developing a new nuclear medicine imaging technique for measuring liquid absorption in the airways that can be applied to screen new medications being developed to treat cystic fibrosis (CF). The investigators believe that the absorption of the small molecule radiopharmaceutical Indium 111 diethylene triamine pentaacetic acid (In-DTPA) will indicate changes in liquid absorption in the airways and demonstrate whether new CF medications will be effective. In this study the investigators will determine whether the imaging technique will demonstrate similar results when it is repeated on different days. They will also determine how their results change when subjects utilize several common CF medications.

DETAILED DESCRIPTION:
Cystic Fibrosis (CF) is an autosomal recessive genetic disease, caused by mutations of the Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) that impairs ion transport at epithelial surfaces. This results in the accumulation of dehydrated secretions in the airways and chronic infection and inflammation in the lungs, leading to significant morbidity and mortality. The investigators understanding of CF pathogenesis has increased substantially and many new targeted therapies are being developed to treat this disease, however, the measurements of clinical efficacy used to evaluate these therapies require long trials to demonstrate an effect. New translational techniques are needed to assess changes in the most basic aspects of the disease and allow for the rapid screening of disease-altering therapies. The investigators have recently developed a novel aerosol-based imaging technique to measure liquid absorption in the airways - a central pathophysiological process related to CFTR dysfunction. The investigators propose that airway liquid hyper-absorption is a key link between cellular defects in ion and fluid transport and progressive airway dysfunction in CF. Thus The investigators technique may provide a measure of disease severity and rapid indication of therapeutic correction in advance of currently available outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* subjects 18 years old or older with a diagnosis of cystic fibrosis as determined by sweat test or genotype and clinical symptoms who are clinically stable as determined by a physician co-investigator

Exclusion Criteria:

* one second forced expiratory volume (FEV1) <50% of predicted
* nursing mother
* positive urine pregnancy test or unwilling to test
* cigarette smoker
* unwilling to stop hypertonic saline therapy for 72 hours prior to each test day
* are intolerant to hypertonic saline (response only)
* are intolerant to any inhaled therapies (response only)
* fail mannitol tolerance testing (response only)
* have a history of excessive (uncontrollable) coughing after an osmotic stimulus (response only)
* have a history of hemoptysis (response only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
absorptive clearance variability | 30 days
  The difference in absorptive clearance measured on two different study days in the same subjects as an indicator of measurement variability
absorptive clearance response | 14 day
  The change in absorptive clearance demonstrated in response to therapy when compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Tim Corcoran, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Corcoran TE, Thomas KM, Brown S, Myerburg MM, Locke LW, Pilewski JM. Liquid hyper-absorption as a cause of increased DTPA clearance in the cystic fibrosis airway. EJNMMI Res. 2013 Feb 27;3(1):14. doi: 10.1186/2191-219X-3-14. PMID 23446051
- [Background] Corcoran TE, Thomas KM, Myerburg MM, Muthukrishnan A, Weber L, Frizzell R, Pilewski JM. Absorptive clearance of DTPA as an aerosol-based biomarker in the cystic fibrosis airway. Eur Respir J. 2010 Apr;35(4):781-6. doi: 10.1183/09031936.00059009. Epub 2009 Aug 28. PMID 19717485
- [Derived] Locke LW, Myerburg MM, Weiner DJ, Markovetz MR, Parker RS, Muthukrishnan A, Weber L, Czachowski MR, Lacy RT, Pilewski JM, Corcoran TE. Pseudomonas infection and mucociliary and absorptive clearance in the cystic fibrosis lung. Eur Respir J. 2016 May;47(5):1392-401. doi: 10.1183/13993003.01880-2015. Epub 2016 Mar 23. PMID 27009167